CLINICAL TRIAL: NCT01063517
Title: A Randomised, Double Blinded, Multicentre Phase II Study to Assess the Efficacy of Olaparib (AZD2281, KU-0059436) in Combination With Paclitaxel Versus Paclitaxel in Patients With Recurrent or Metastatic Gastric Cancer Who Progress Following First-line Therapy
Brief Title: Efficacy Study of Olaparib With Paclitaxel Versus Paclitaxel in Gastric Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0810C00039
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
Keywords: Poly(ADP ribose); polymerase (PARP); Gastric cancer; olaparib; PARP inhibitor; ATM AZD2281; Ku0059436; Homologous Recombination deficiency (HRD); Recurrent gastric cancer; metastatic gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — olaparib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Olaparib + paclitaxel
  Interventions: Drug: olaparib; Drug: paclitaxel
- 2 (Active Comparator): paclitaxel + placebo
  Interventions: Drug: paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: olaparib — 100mg BID oral tablet continuous
  Arms: 1
Drug: paclitaxel — iv infusion 80mg/m2 on Day 1, 8 and 15 of a 28 day cycle
  Other Names: Taxol
Drug: Placebo — 100mg BID oral tablet to match olaparib tablet
  Arms: 2

SUMMARY:
To assess the efficacy of olaparib when given in combination with paclitaxel compared with paclitaxel alone as defined by progression-free survival (PFS), in all patients with recurrent and metastatic gastric cancer who progress following first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic gastric cancer that has progressed following first line-therapy
* Confirmed ATM protein status by IHC archival tumour sample
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed by imaging (CT/MRI) at baseline and follow up visits

Exclusion Criteria:

* More than one prior chemotherapy regimen for the treatment of gastric cancer in the metastatic or recurrent setting
* Any previous treatment with a PARP inhibitor, including olaparib
* Patients with second primary cancer, except; adequately treated non melanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for >5 years

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2012-05-11 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Yung-Jue Bang, MD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Jeonnam
  - Research Site, Seoul
  - Research Site, Taegu

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Chan KH, Rutazanaa D, Wray C, Thosani N, Yang V, Cen P. Promising Response of Olaparib in Patient With Germline ATM-Mutated Metastatic Gastric Cancer. J Investig Med High Impact Case Rep. 2024 Jan-Dec;12:23247096241240176. doi: 10.1177/23247096241240176. PMID 38504422
- See also: CSR_Synopsis_D0810C00039 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1677&filename=D0810C00039.pdf
- See also: D0810C00039Protocol_and_Amendments_redacted_SECURE — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1677&filename=D0810C00039Protocol_and_Amendments_redacted_SECURED.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 sites in South Korea. Enrolment started in February 2010 and was completed in May 2012. In total 124 patients were randomised in the study (62 in the olaparib+paclitaxel arm and 62 in the placebo+paclitaxel arm).
Pre-assignment Details: Patients of either sex, age more than 17 years with recurrent or metastatic gastric cancer that had progressed following first line therapy, a confirmed Ataxia Telangiectasia Mutation (ATM) status, Eastern Co operative Oncology Group (ECOG) performance status ≤2, normal organ and bone marrow function, and life expectancy ≥16 weeks.
Groups:
- Olaparib+Paclitaxel: Olaparib 100 mg twice daily in tablet formulation in combination with paclitaxel 80 mg/m2 intravenous on Days 1, 8, and 15 of a 4 week schedule. It was expected that patients would receive between 6 to 10 cycles of paclitaxel after which olaparib dose was increased to 200 mg bd as monotherapy.
- Placebo+Paclitaxel: Matching placebo 100 mg twice daily in tablet formulation in combination with paclitaxel 80 mg/m2 intravenous on Days 1, 8, and 15 of a 4 week schedule. It was expected that patients would receive between 6 to 10 cycles of paclitaxel after which placebo dose was increased to 200 mg bd as monotherapy.
Period: Overall Study
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Started | 62 | 62
Received Randomised Treatment | 61 | 62
Completed | 4 | 2
Not Completed | 58 | 60
Not completed — Consent withdrawal | 1 | 0
Not completed — Study reached data cut-off | 19 | 7
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 33 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of randomisation
  years | 59.0 (11.61) | 59.4 (11.98) | 59.2 (11.75)
Age, Customized [Number; unit: Participants] — Age category
  Participants
    < 50 years | 13 | 10 | 23
    >=50 to <65 years | 22 | 30 | 52
    >= 65 years | 27 | 22 | 49
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 13 | 18 | 31
    Male | 49 | 44 | 93
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Asian | 62 | 62 | 124
    Other | 0 | 0 | 0
ATM status [Number; unit: Participants] — Ataxia-Telangiectasia Mutation (ATM) protein testing
  Participants
    Negative | 31 | 32 | 63
    Positive | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in the Overall Study Population
Description: PFS is defined as the time from randomisation till objective progression or death. In absence of progression or death, the time is calculated from randomisation till last evaluable scanning visit.
Time Frame: Tumour assessments were carried out at baseline and then follow up assessments taken every 8 weeks up to Week 40 and then every 16 weeks until objective disease progression as defined by RECIST 1.1, assessed maximum up to 27 months
Population: Full analysis set including all randomised patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 62 | 62
months | 3.91 [3.02 to 7.13] | 3.55 [1.74 to 5.82]
Statistical Analysis 1: Comparison: Olaparib+Paclitaxel vs Placebo+Paclitaxel; The analysis was performed using a Cox proportional hazards model with factors for treatment group, ATM status and gastrectomy (full, partial, none); Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 80% CI 2-sided [0.62 to 1.03] — The numerator of the hazard ratio is hazards of progression in olaparib+paclitaxel group and denominator is hazards of progression in placebo+paclitaxel group. Confidence intervals are calculated using the profile-likelihood method

2. Primary Outcome: Progression Free Survival (PFS) in Patients With Tumours Defined as Homologous Recombination Deficient by Loss of Ataxia-Telangiectasia Mutation (ATM) Protein [ATM Negative Patients]
Description: as for outcome 1
Time Frame: Tumour assessments are carried out at baseline and then follow up assessments taken every 8 weeks up to Week 40 and then every 16 weeks until objective disease progression as defined by RECIST 1.1, assessed maximum up to 27 months
Population: Full analysis set including randomised ATM negative patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 31 | 32
months | 5.29 [3.38 to 5.72] | 3.68 [1.77 to 5.82]
Statistical Analysis 1: Comparison: Olaparib+Paclitaxel vs Placebo+Paclitaxel; The analysis was performed using a Cox proportional hazards model with factors for treatment group and gastrectomy (full, partial, none); Test type: Superiority or Other; Hazard Ratio (HR) = 0.74, 80% CI 2-sided [0.51 to 1.08] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival (OS) in the Overall Study Population
Description: Overall survival is defined as the duration from randomisation till death. In absence of death, the time is calculated from randomisation till the date subject last known to be alive.
Time Frame: Survival follow up from randomisation till death of the patient or till end of study in absence of death, assessed maximum up to 27 months
Population: Full analysis set including all randomised patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 62 | 62
months | 13.1 [7.10 to NA] — NA: There were insufficient events to calculate. | 8.3 [5.30 to 14.90]
Statistical Analysis 1: Comparison: Olaparib+Paclitaxel vs Placebo+Paclitaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.56, 80% CI 2-sided [0.41 to 0.75] — The numerator of the hazard ratio is hazards of death in olaparib+paclitaxel group and denominator is hazards of death in placebo+paclitaxel group. Confidence intervals are calculated using the profile-likelihood method

4. Secondary Outcome: Overall Survival (OS) in ATM Negative Patients
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Full analysis set including randomised ATM negative patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 31 | 32
months | NA [9.30 to NA] — More than 50% of patients were alive at the data cut-off date | 8.20 [5.10 to 13.10]
Statistical Analysis 1: Comparison: Olaparib+Paclitaxel vs Placebo+Paclitaxel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.35, 80% CI 2-sided [0.22 to 0.56] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Objective Response Rate (ORR) in the Overall Study Population
Description: Objective response rate is the proportion of patients with at least one measurable lesion at baseline, who experienced complete or partial response at least once during the assessment period, according to the definitions of Response Evaluation Criteria In Solid Tumours (RECIST version 1.1).
Time Frame: Tumour assessments carried out at baseline, 28 days before randomisation then every 8 weeks until week 40, after week 40 assessments will be carried out every 16 weeks until objective disease progression, assessed maximum up to 27 months
Population: Evaluable for response population - randomised patients having measurable disease at baseline.
Measure: Number; unit: Participants
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 53 | 47
Participants | 14 | 9

6. Secondary Outcome: Objective Response Rate (ORR) in the ATM Negative Patients
Description: Objective response rate is the proportion of ATM negative patients with at least one measurable lesion at baseline, who experienced complete or partial response at least once during the assessment period, according to the definitions of Response Evaluation Criteria In Solid Tumours (RECIST version 1.1).
Time Frame: as for outcome 5
Population: Evaluable for response population ATM negative patients - randomised ATM negative patients having measurable disease at baseline.
Measure: Number; unit: Participants
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 26 | 23
Participants | 9 | 6

7. Secondary Outcome: Percentage Change in Tumour Size at Week 8 in the Overall Study Population
Description: Percentage change in tumour size from baseline to Week 8 calculated as 100 X (week 8 tumour size - baseline tumour size) / (baseline tumour size)
Time Frame: Tumour scans done at Baseline and week 8
Population: Evaluable for response population - randomised patients having measurable disease at baseline.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 52 | 47
Percent change | -5.8 (29.09) | 2.2 (35.6)

8. Secondary Outcome: Percentage Change in Tumour Size at Week 8 in the ATM Negative Patients
Description: as for outcome 7
Time Frame: Tumour scans done at Baseline and week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 26 | 23
Percent change | -6.9 (29.31) | -5.9 (26.36)

9. Secondary Outcome: Time to Deterioration in Global Quality of Life (QoL) Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of Global QoL score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: Questionnaire data collected at Baseline ie on or before date of randomisation, every 4 weeks post baseline, assessed maximum up to 27 months
Population: Randomised patients having global score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 3.6 (29.31) [1.1 to 8.3] | 2.8 (26.36) [1.8 to 5.7]

10. Secondary Outcome: Time to Deterioration in QoL Fatigue Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of fatigue score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having fatigue score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 1.9 (29.31) [0.9 to NA] — NA: There were insufficient events to calculate. | 1.8 (26.36) [0.9 to 5.1]

11. Secondary Outcome: Time to Deterioration in QoL Nausea & Vomiting Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of nausea & vomiting domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having nausea & vomiting domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 3.7 (29.31) [1.65 to 13.9] | 3.7 (26.36) [1.8 to 7.6]

12. Secondary Outcome: Time to Deterioration in QoL Pain Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of pain domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having pain domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 3.2 (29.31) [1.8 to 5.5] | 3.1 (26.36) [1.0 to 5.7]

13. Secondary Outcome: Time to Deterioration in QoL Dysphagia Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of dysphagia domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having dysphagia domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 3.7 (29.31) [2.2 to 12.6] | 1.9 (26.36) [0.9 to 6.4]

14. Secondary Outcome: Time to Deterioration in QoL Eating Restriction Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of eating restriction domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having eating restriction domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 4.6 (29.31) [2.5 to 12.9] | 5.1 (26.36) [2.2 to 8.9]

15. Secondary Outcome: Time to Deterioration in QoL Stomach Pain Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of stomach pain domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having stomach pain domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 6.9 (29.31) [3.7 to NA] — NA: There were insufficient events to calculate. | 5.7 (26.36) [2.8 to 9.2]

16. Secondary Outcome: Time to Deterioration in QoL Reflux Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of reflux domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having reflux domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 4.3 (29.31) [2.1 to 13.9] | 2.8 (26.36) [1.0 to 5.7]

17. Secondary Outcome: Time to Deterioration in QoL Anxiety Domain Score in the Overall Study Population
Description: Time calculated from randomisation till worsening of anxiety domain score based on European Organisation for Research and Treatment of Cancer (EORTC) questionnaire data
Time Frame: as for outcome 9
Population: Randomised patients having anxiety domain score calculated at baseline and at least one post baseline visit
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Olaparib+Paclitaxel | Placebo+Paclitaxel
Number analyzed (Participants) | 61 | 60
months | 2.8 (29.31) [1.1 to 12.2] | 1.9 (26.36) [1.0 to 5.1]

ADVERSE EVENTS:
Arm/Group | OLAPARIB 100MG BD + PACLITAXEL / OLAPARIB 200MG BD | PLACEBO 100MG BD + PACLITAXEL / PLACEBO 200MG BD
Serious Adverse Events (participants affected / at risk) | 17/61 | 23/62
Other Adverse Events (participants affected / at risk) | 61/61 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLAPARIB 100MG BD + PACLITAXEL / OLAPARIB 200MG BD (N=61) | PLACEBO 100MG BD + PACLITAXEL / PLACEBO 200MG BD (N=62)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 2 (2)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 2 (2)
PAIN (General disorders) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 1 (1) | 2 (2)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
ALCOHOLISM (Psychiatric disorders) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLAPARIB 100MG BD + PACLITAXEL / OLAPARIB 200MG BD (N=61) | PLACEBO 100MG BD + PACLITAXEL / PLACEBO 200MG BD (N=62)
ANAEMIA (Blood and lymphatic system disorders) | 11 (17) | 12 (23)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 46 (162) | 40 (127)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 2 (2)
EYE PAIN (Eye disorders) | 1 (1) | 1 (1)
PTERYGIUM (Eye disorders) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 (4) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 (4) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 (18) | 16 (19)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 (9) | 8 (10)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
BREATH ODOUR (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 20 (34) | 17 (28)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 11 (16) | 10 (13)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
ERUCTATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
GINGIVITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
LIP PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 21 (26) | 26 (32)
ORAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0)
REFLUX GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 3 (6)
TOOTHACHE (Gastrointestinal disorders) | 3 (3) | 1 (1)
VOMITING (Gastrointestinal disorders) | 9 (11) | 14 (16)
CHILLS (General disorders) | 1 (1) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 15 (15) | 19 (24)
GENERALISED OEDEMA (General disorders) | 0 (0) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (5) | 3 (3)
IRRITABILITY (General disorders) | 0 (0) | 2 (2)
LOCALISED OEDEMA (General disorders) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 4 (4) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (2)
OEDEMA (General disorders) | 1 (1) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 6 (7)
PAIN (General disorders) | 3 (3) | 2 (2)
PYREXIA (General disorders) | 6 (7) | 13 (16)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 2 (2)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (5) | 4 (7)
PHARYNGITIS (Infections and infestations) | 1 (1) | 2 (2)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1)
RHINITIS (Infections and infestations) | 1 (1) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (9) | 5 (5)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (6) | 4 (5)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (4) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 (3) | 5 (5)
HAEMOGLOBIN (Investigations) | 0 (0) | 1 (3)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (11) | 1 (1)
WEIGHT DECREASED (Investigations) | 4 (4) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 23 (30) | 25 (34)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (8)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 (17) | 22 (32)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 11 (12) | 7 (14)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2)
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 22 (22) | 13 (15)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 8 (8) | 10 (11)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (2)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERED (Psychiatric disorders) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 3 (3) | 5 (5)
HAEMOGLOBINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
MICTURITION URGENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRAL PAIN (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
GENITAL RASH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC DISCOMFORT (Reproductive system and breast disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (8)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (13)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
TONSILLAR INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 30 (30) | 29 (29)
BLISTER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (11) | 3 (4)
RASH (Skin and subcutaneous tissue disorders) | 8 (10) | 8 (11)
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
PERIPHERAL COLDNESS (Vascular disorders) | 0 (0) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 14 (15) | 10 (11)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 19 (29) | 15 (22)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 2 (2)
FURUNCLE (Infections and infestations) | 1 (1) | 0 (0)
HERPES VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5) | 4 (6)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3) | 4 (5)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (3)
INSOMNIA (Psychiatric disorders) | 7 (8) | 4 (6)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less